CLINICAL TRIAL: NCT03401762
Title: Wearable MCI to Reduce Muscle Co-activation in Acute and Chronic Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Shirley Ryan AbilityLab (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Marc Slutzky, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00203644
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Stroke; Stroke, Acute
Keywords: rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded as to sham vs. intervention, but not as to which interventional arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Chronic stroke MCI Electromyogram (EMG) pairs (Experimental): Decoupling 2 muscles at a time with MCI
  Interventions: Behavioral: MCI
- Chronic stroke MCI EMG triplets (Experimental): Decoupling 3 muscles at a time with MCI
  Interventions: Behavioral: MCI
- Chronic stroke MCI while reaching (Experimental): Decoupling muscles with MCI while reaching to targets
  Interventions: Behavioral: MCI
- Chronic stroke Sham MCI (Sham Comparator): Sham control group
  Interventions: Behavioral: Sham MCI
- Acute stroke MCI (Experimental): Decoupling muscles with MCI in acute stroke subjects
  Interventions: Behavioral: MCI
- Acute stroke Sham MCI (Sham Comparator): Acute stroke subjects sham comparator
  Interventions: Behavioral: Sham MCI

INTERVENTIONS:
Behavioral: MCI — EMG-controlled game
  Arms: Acute stroke MCI; Chronic stroke MCI EMG triplets; Chronic stroke MCI Electromyogram (EMG) pairs; Chronic stroke MCI while reaching
Behavioral: Sham MCI — Sham control game
  Arms: Acute stroke Sham MCI; Chronic stroke Sham MCI

SUMMARY:
The purpose of the study is to explore the feasibility of using a wearable device, called a myoelectric-computer interface (MCI), to improve arm movement in people who have had a stroke.

Impaired arm movement after stroke is caused not just by weakness, but also by impaired coordination between joints due to abnormal co-activation of muscles. These abnormal co-activation patterns are thought to be due to abnormal movement planning.The MCI aims to reduce abnormal co-activation by providing feedback about individual muscle activations.

This randomized, controlled, blinded study will test the home use of an MCI in chronic and acute stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

Chronic stroke participants

* Hemiparesis from first ever stroke at least 6 months prior to screening
* Severe motor impairment (FMA of 7-30)
* At least some voluntary shoulder and elbow muscle activation.

Acute stroke participants

* Hemiparesis from first ever stroke within the past 21 days
* Severe motor impairment (FMA of 3-20), or total Manual Motor Score of 1-8 combined in Shoulder Abduction and Finger Extensors

Exclusion Criteria:

* Cognitive impairment with at least moderately impaired attention, or unable to follow instructions of the MCI task
* Visual impairment (such as hemianopia) preventing full view of the screen
* Anesthesia or neglect in the affected arm, or visual hemineglect (score of 2 on the NIH Stroke Scale Extinction and Inattention subtest).
* Participation in another study on the affected arm within 6 weeks of enrollment or any pharmacological study
* Inability to understand or follow commands in English due to aphasia or other reason
* Diffuse or multifocal infarcts
* Substantial arm pain preventing participation for 90 minutes a day
* New spasticity treatment (pharmacological or Botox)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2018-01-15 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Wolf Motor Function Test | baseline to 6 weeks
  Timed

SECONDARY OUTCOMES:
Fugl-Meyer Assessment - Upper Extremity (UE) | baseline to 6 weeks
Motor Activity Log | baseline to 6 weeks
Modified Ashworth Scale | baseline to 6 weeks
  Total score
Fugl-Meyer Assessment UE | baseline to 10 weeks
Wolf Motor Function Test | baseline to 10 weeks
  Timed

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Khorasani A, Gorski CM, Hung NT, Hulsizer J, Paul V, Tomic G, Prakash PR, Park S, Seo G, Houskamp EJ, Lanis J, Hunzeker M, King E, Chappel A, Jampol A, Patel P, Gallagher C, Galant R, Rucker G, Lee J, Harvey R, Roh J, Slutzky MW. Wearable Myoelectric Interface for Neurorehabilitation (MINT) to Recover Arm Function: a Randomized Controlled Trial. medRxiv [Preprint]. 2025 Jun 25:2025.06.24.25330240. doi: 10.1101/2025.06.24.25330240. PMID 40666333
- [Derived] Khorasani A, Hulsizer J, Paul V, Gorski C, Dhaher YY, Slutzky MW. Myoelectric interface for neurorehabilitation conditioning to reduce abnormal leg co-activation after stroke: a pilot study. J Neuroeng Rehabil. 2024 Jan 20;21(1):11. doi: 10.1186/s12984-024-01305-0. PMID 38245730
- [Derived] Khorasani A, Hulsizer J, Paul V, Gorski C, Dhaher YY, Slutzky MW. Myoelectric interface for neurorehabilitation conditioning to reduce abnormal leg co-activation after stroke: a pilot study. Res Sq [Preprint]. 2023 Oct 9:rs.3.rs-3398815. doi: 10.21203/rs.3.rs-3398815/v1. PMID 37886579
- [Derived] Hung NT, Paul V, Prakash P, Kovach T, Tacy G, Tomic G, Park S, Jacobson T, Jampol A, Patel P, Chappel A, King E, Slutzky MW. Wearable myoelectric interface enables high-dose, home-based training in severely impaired chronic stroke survivors. Ann Clin Transl Neurol. 2021 Sep;8(9):1895-1905. doi: 10.1002/acn3.51442. Epub 2021 Aug 20. PMID 34415114